CLINICAL TRIAL: NCT01846936
Title: A Randomized, Prospective Trial Comparing Double-lumen Tube and Bronchial Blocker With or Without Modified Disconnection Technique
Brief Title: Disconnection Technique With a Bronchial Blocker for Improving Lung Deflation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Sung Yong Park, associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AJIRB-DEV-DE1012-001
Record Dates: First submitted 2012-10-24; First posted 2013-05-06 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Pneumothorax
Keywords: one lung ventilation; efficacy; bronchial blocker
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- DLT with conventional technique (Experimental): The double lumen tube is introduced into the glottis under direct laryngoscopy. After the bronchial cuff had passes the vocal cords, the tube is rotated counterclockwise 90° and advanced until a slight resistance was encountered.
  One lung ventilation is initiated after the lumen of operative lung is clamped and opened.
  Interventions: Procedure: DLT with conventional technique
- BB with conventional technique (Active Comparator): The brochial blocker (BB) is introduced through the endotracheal tube to the desired bronchus under fiberoptic bronchoscopy (FOB) vision by turning the device's steering wheel.
  The BB cuff is inflated with air under FOB vision with the volume necessary to seal the bronchus and initiate one lung ventilation. And then, dependent lung is ventilated.
  Interventions: Procedure: BB with conventional technique
- Disconnection technique (Active Comparator): Disconnection technique; 1) before initiating OLV, we turned-off the ventilator and fully opened the adjustable pressure limiting valve allowing both lungs to collapse, and 2) after loss of the carbon dioxide trace on the capnograph, 3) inflated the BB cuff with air, and 4) turned-on the ventilator allowing only dependent-lung reventilation.
  Interventions: Procedure: Disconnection technique

INTERVENTIONS:
Procedure: DLT with conventional technique — The double lumen tube is introduced into the glottis under direct laryngoscopy. After the bronchial cuff had passes the vocal cords, the tube is rotated counterclockwise 90° and advanced until a slight resistance was encountered.
  Arms: DLT with conventional technique
Procedure: BB with conventional technique — The brochial blocker (BB) is introduced through the endotracheal tube to the desired bronchus under FOB vision by turning the device's steering wheel.
  The BB cuff is inflated with air under FOB vision with the volume necessary to seal the bronchus and initiate one lung ventilation.
  Arms: BB with conventional technique
Procedure: Disconnection technique — Disconnection technique 1) deflate of the blocker cuff, 2) turn-off the ventilator and opened the APL valve allowing both lungs to collapse, 3) after loss of carbon dioxide trace in the capnograph, reinflate blocker cuff with the same volume of air as during the initial insertion, 4) reconnect the tube to the ventilator allowing only dependent-lung reventilation with a 5 cmH2O positive end-expiratory pressure preceded by a single recruitment maneuver performed by elevating the airway pressure to 40 cmH2O for 7 seconds.
  Arms: Disconnection technique

SUMMARY:
One lung ventilation (OLV) is accomplished with a double lumen tube (DLT) or a bronchial blocker (BB). In this study, the investigators compared the effectiveness of lung collapse using DLT, BB with spontaneous collapse, and BB with disconnection technique.

DETAILED DESCRIPTION:
In selecting this maneuver of OLV, lung collapse is a major concern because it permits adequate surgical exposure. Although once lung deflation was achieved, the overall clinical performance appears to be similar, BB takes longer to deflate the operative lung and there is some conflict reports as to BB provides a similar degree of lung deflation compared to that of DLT.

The aim of this study was to compare the efficacy of BB and DLT for achieving lung collapse, and to evaluate the efficacy of disconnection technique with monitoring the carbon dioxide trace on a capnograph in BB. The investigators further evaluated the disconnection time, which is the time to loss of carbon dioxide trace on the capnograph, needed to facilitate lung collapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic surgery for which OLV is required

Exclusion Criteria:

* Patients with an anticipated difficult intubation with infectious or bleeding lung lesions are excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of three lung isolation methods | Five min from the start of one lung ventilation
  The degree of lung collapse after 5 min from the start of OLV. The degree of lung collapse was assessed using a lung collapse score (0 = no collapse, to 10 = complete collapse) by one thoracic surgeon. The surgeon who assessed the lung collapse was absent from the operating room during DLT or BB placement and was blinded to the airway device.
Effectiveness of three lung isolation methods | Ten min from the start of one lung ventilation
  The degree of lung collapse after 5 min from the start of OLV. The degree of lung collapse was assessed using a lung collapse score (0 = no collapse, to 10 = complete collapse) by one thoracic surgeon. The surgeon who assessed the lung collapse was absent from the operating room during DLT or BB placement and was blinded to the airway device.

SECONDARY OUTCOMES:
The disconnection time | The time to loss the carbon dioxide trace on the capnograph (30 seconds)
  Before initiating OLV in group 3, we turned-off the ventilator and fully opened the adjustable pressure limiting valve allowing both lungs to collapse. And then, the time which capnograph lose the carbon dioxide curve is considered the disconnection time required for both lungs to collapse before initiating one lung ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Park, MD, Principal Investigator — Ajou University
Locations (1):
- Ajou University Hospital, Suwon, Gyung Gi, South Korea